CLINICAL TRIAL: NCT02216981
Title: A Pilot Randomised Controlled Trial to Assess the Feasibility of Cognitive Behavioural Therapy (CBT) Delivered in Time-Intensive and Weekly Treatment Formats for Treatment Resistant Obsessive Compulsive Disorder (OCD).
Brief Title: Examining the Feasibility and Acceptability of Good Quality Intensive CBT for OCD and Good Quality Weekly CBT for OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bath (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); Avon and Wiltshire Mental Health Partnership NHS Trust (Other Government)
Responsible Party: Principal Investigator, Josie Millar, Lecturer & Clinical Psychologist, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MILSALK1
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Obsessive Compulsive Disorder (OCD); Cognitive Behavioural Therapy (CBT); Intensive therapy; Intensive treatment; Treatment Resistant
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensive Cognitive Behavioural Therapy (Experimental): Intensive CBT (an average of 12-18 hours of CBT offered in an intensive format, delivered on 2-3 days per week over a period of 3 weeks)
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Weekly Cognitive Behavioural Therapy (Active Comparator): Weekly CBT (an average of 12-18 hours of CBT delivered in 60-90 minute sessions on a weekly basis)
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Wait list (No Intervention): Wait list (3 months). Participants randomized to wait list will commence treatment after 3 months, in the treatment condition to which they are re-randomized (either Intensive or Weekly CBT).

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT)
  Arms: Intensive Cognitive Behavioural Therapy; Weekly Cognitive Behavioural Therapy

SUMMARY:
The purpose of this study is to examine how feasible and acceptable it is to deliver a talking treatment called Cognitive Behavioural Therapy (CBT) in two different formats for people who have had treatment for OCD in the past but it didn't work out for them.

The two different treatment formats are CBT delivered on a weekly basis (which is approximately 12-18 hours of therapy delivered weekly for 60-90 minutes each session, followed by 1-3 monthly follow up sessions as needed) and CBT offered in an intensive format (which is having approximately 12-18 hours of therapy all in a 3-week period, followed by 1-3 monthly follow up sessions as needed).

DETAILED DESCRIPTION:
The main aim of this study is to assess the feasibility and acceptability of Intensive CBT for treatment resistant OCD when participants are randomized to this format.

This study aims to establish an estimate of the relative efficacy of both Intensive and Weekly CBT when compared individually to wait list, for participants with a diagnosis of OCD, who have previously not responded to CBT.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of OCD (as confirmed by the administration of the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 4th ed.) (DSM-IV) (SCID-I) .
* Participant identifies their main problem as OCD.
* Participant has not responded to one or more trials CBT
* Yale-Brown Obsessive Compulsive Scale (YBOCS) score of 16 or above.
* No change in psychotropic medication (if applicable) for at least 8 weeks prior to study entry. (If such a change has taken place there will be an option for the participant to take part once the medication has been stabilised).
* No intention to change psychotropic medication during the course of the trial
* Able to speak and read every day English

Exclusion Criteria:

* Severe psychiatric problem that requires separate treatment at an immediate basis and is linked to risk.
* Drug and/or alcohol dependence in last three months
* History of Psychosis or Bipolar Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Yale- Brown Obsessive Compulsive Scale (Y-BOCS) & Obsessive Compulsive Inventory | Assessment, end of treatment (at 3 weeks for Intensive & 12-15 weeks for weekly treatment) and follow up (at 3 & 6 months post treatment completion for both groups).
  The Y-BOCS is Clinician administered and the OCI is self report, both measures assess the severity of OCD symptoms.
  These measures will be used to assess change in symptom severity from base line to end of treatment and to assess if there has been a change at end of treatment, if this is maintained at 3 and 6 months following the completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Josie FA Millar, Principal Investigator — University of Bath; Paul M Salkovskis, Study Director — University of Bath
Locations (2):
- United Kingdom (2):
  - Centre for Specialist Psychological Treatments of Anxiety and Related Problems (CSPTARP), Bath, Bath
  - Centre for Anxiety Disorders and Trauma (CADAT), London, Denmark Hill